CLINICAL TRIAL: NCT01124708
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter, Fixed Dose Titration Study to Assess Efficacy, Safety, and Tolerability of TC-5619 in Adults With Attention Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Efficacy, Safety, and Tolerability of TC-5619 in Adults With Attention Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TC-5619-238-CRD-002; PRO-05619-CRD-002
Record Dates: First submitted 2010-05-05; First posted 2010-05-17 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2011-10

CONDITIONS: ADHD
Keywords: ADHD; Attention Deficit Hyperactive Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be provided as white, opaque gelatin capsules in sham strengths of 1mg, 5mg, and 25mg
  Interventions: Drug: Placebo
- TC-5619 (Active Comparator): TC-5619-238 will be provided as white, opaque gelatin capsules in strengths of 1mg, 5mg, and 25mg (as free base). Subjects will take 1mg TC-5619, 5mg TC-5619, 25mg TC-5619, one capsule once daily p.o.
  Interventions: Drug: TC-5619-238

INTERVENTIONS:
Drug: TC-5619-238 — TC-5619-238 will be provided as white, opaque gelatin capsules in strengths of 1mg, 5mg, and 25mg (as free base). Subjects will take 1mg TC-5619, 5mg TC-5619, 25mg TC-5619, or matching placebo - one capsule once daily p.o.
  Arms: TC-5619
Drug: Placebo — Placebo will be provided as white, opaque gelatin capsules in sham strengths of 1mg, 5mg, and 25mg
  Arms: Placebo

SUMMARY:
ADHD has been associated with persistent deficits in the efficient allocation of attention and supports the notion that regulation of the cholinergic system may improve these cognitive deficits in ADHD. It has been suggested that the effects of nicotine are most pronounced on tasks that demand effortful processing (Rusted and Warburton 1994). In addition, a recent theory proposes that the cholinergic system allocates additional attentional resources during tasks that are demanding (i.e. sustained attention, set shifting, etc; Sarter and Bruno 1997). Thus it may be that in ADHD, cholinergic systems are under-responsive or under-developed and thus stimulation of nicotinic receptors via nicotinic agents may result in improved cognitive performance particularly on tests requiring effortful processing.

DETAILED DESCRIPTION:
A randomized, parallel, forced-titration design is being used to assess effects of TC-5619 versus placebo on efficacy. A parallel group design allows the effects of TC-5619 to be clearly established, and the randomized nature of the design allows minimization of observer and subject bias. Because a forced dose up-titration design will be used, effects of individual doses will be preliminary, because the design confounds dose with time.

The doses chosen (1mg, 5mg, and 25mg) reflect an appropriate range around the anticipated efficacious dose (3-10 mg), based upon preclinical extrapolations to the human, and upon the pro-cognitive effects of TC-5619 identified by CDR in the MRD study (Targacept Study TC-5619-238-CLP-002).

All subjects will be tobacco non-users. It is possible that tobacco (nicotine) interferes with α7 NNR-mediated effects.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ADHD per DSM-IV TR criteria
2. Score > 2 on at least 6 of 9 items in at least 1 subscale of the CAARS-INV
3. Score > 4 (at least moderate) on the Clinical Global Impression-Severity (CGI-S) index
4. Age 18 - 65, male or female
5. Tobacco non-users as indicated by lack of tobacco use within the last year prior to Screening, and by negative urinary cotinine level of < 50ng/mL after quantification
6. Able to understand and sign informed consent

Exclusion Criteria:

1. Current DSM-IV Axis I psychiatric disorder other than ADHD; use of MINI to exclude other major DSM-IV TR psychiatric diagnoses
2. Known or suspected drug abuse within the last 12 months prior to Screening
3. Urine drug screen positive for illegal or non-prescribed drugs at Screening
4. Patients at imminent risk of suicide or of danger to themselves or others
5. Use of drugs affecting cognitive function within 3 weeks prior to Day 1, including use of any medications for treatment of ADHD. Any medication wash-outs must be completed during the 3 weeks between Screening and Day 1.
6. Any other restricted or prohibited drugs.
7. Other concomitant medications that have been changed within 4 weeks prior to Screening
8. Unable to comply with study procedures in opinion of investigator, including CogState ADHD test battery
9. History of significant other major or unstable neurological, metabolic, hepatic, renal, hematological, pulmonary, CV, GI, or urological disorder; or diagnosis of major depressive disorder
10. Myocardial infarction within past year
11. Seizure disorder within past year
12. Type 1 diabetes mellitus (DM); type 2 DM that requires medication (diet-controlled allowed)
13. HbA1C > 7.4 at Screening
14. BMI < 15 or > 35; male weight < 100 lbs; female weight < 80 lbs.
15. Current TB or known systemic infection (HBV, HCV, HIV)
16. Clinically significant finding on physical exam
17. Clinically significant lab or ECG abnormality that could be a safety issue in the study, including QTcF > 450 (males) or QTcF > 480msec (females), and excluding LFTs > 1.5 times upper limits of normal
18. Women of child-bearing potential and men unwilling or unable to use accepted methods of birth control
19. Women with a positive pregnancy test, or who are lactating
20. Participation in another clinical trial in last 3 months prior to Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
CAARS-INV ADHD-rating scale | Week 12
  •Clinician-administered ADHD-rating scale (CAARS-INV) and is the total of 3 subscales: Inattention, Hyperactivity-Impulsivity, and ADHD Index [ Time Frame: Week -3, Day 1, Week 1, Week 4 (evaluation of 1mg dose); Week 8 (evaluation of 5mg Dose); and Week 12 (evaluation of 25mg dose)]

SECONDARY OUTCOMES:
CAARS-INV subscales | Week 12
  CAARS-INV subscales: Inattention, Hyperactivity-Impulsivity, and ADHD Index, obtained [Time frame: Week -3, Day 1, Week 1, Week 4, Week 8, Week 12,Early Withdrawal (EW)]
CogState ADHD Battery | Week 12
  CogState ADHD test battery [Time frame: Week -3, Day 1, Week 1, Week 4, Week 8, Week 12,Early Withdrawal (EW)]
CogState Stop-Signal Task scores | Week 12
  CogState Stop-Signal Task scores [Time frame: Week -3, Day 1, Week 1, Week 4, Week 8, Week 12,Early Withdrawal (EW)]
CAARS-Self Rating (CAARS-S) total score | Week 12
  CAARS-S total score [Time frame: Week -3, Day 1, Week 1, Week 4, Week 8, Week 12,Early Withdrawal (EW)]

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newhouse, MD, Principal Investigator — Fletcher Allen Health Care, Dept. of Psychiatry
Locations (16):
- United States (16):
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Fidelity Clinical Research, Inc, Lauderhill, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Scientifc Clinical Research, Inc., North Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Atlanta Center For Clinical Research, Atlanta, Georgia
  - CRI Worldwide, LLC (Lourdes Division), Willingboro, New Jersey
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Oregon Center For Clinical Investigations, Inc. (OBBI, Inc.), Portland, Oregon
  - CRI Worldwide, LLC (Kirkbride Division), Philadelphia, Pennsylvania
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Clinical Trials, LP, Austin, Texas
  - Claghorn-Lessem Research Clinic, Houston, Texas
  - Fletch Allen Health Care, Dept. of Psychiatry, Univ. of Vermont, Burlington, Vermont